CLINICAL TRIAL: NCT04992650
Title: Ultrasonic Perfusion Imaging for Monitoring Mastectomy Skin Microcirculation in Post-mastectomy Irradiated Patients Before and After Autologous Fat Transfer
Brief Title: Ultrasonic Perfusion Imaging in Post-mastectomy Irradiated Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-001411; NCI-2021-08914 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-04-01; First posted 2021-08-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Breast Reconstruction; Radiation Dermatitis; Radiation Fibrosis; Fat Grafting
MeSH Terms: conditions — Radiodermatitis; Radiation Fibrosis Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast reconstruction with fat grafting (Experimental): fat grafting
  Interventions: Procedure: Fat grafting
- breast reconstruction without fat grafting (No Intervention): No Fat grafting

INTERVENTIONS:
Procedure: Fat grafting — Fat grafting
  Arms: Breast reconstruction with fat grafting

SUMMARY:
The purpose of this study is to evaluate post-mastectomy breast skin blood supply (perfusion) after radiation therapy, and before and after fat grafting to the breast(s).

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients undergoing immediate tissue expander or implant reconstruction requiring radiation therapy
* Have undergone mastectomy

Exclusion Criteria:

* Patients who are unwilling to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Radiation Fibrosis | 12 months
  Number of subject to experience radiation fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Christin A. Harless, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials